CLINICAL TRIAL: NCT01799551
Title: A Randomised Controlled Trial of Brief Culturally Adapted CBT for Depression in Pakistan
Brief Title: Brief Culturally Adapted Cognitive Behaviour Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Principal Investigator, Fraooq Naeem, President, Pakistan Association of Cognitive Therapists, Pakistan Association of Cognitive Therapists
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PakistanACT
Record Dates: First submitted 2013-02-23; First posted 2013-02-27 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Depression
Keywords: Depression; Culture; CBT; Adaptation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ca CBT (Active Comparator): Experimental arm will receive brief version of Culturally adapted CBT for depression. This is based on our previous work in which we adapted CBT for depression in Pakistan
  Interventions: Behavioral: Ca CBT
- Treatment As Usual (No Intervention): Patients in this arm will get only Treatment As Usual, which normally includes regular follow up and medicines.

INTERVENTIONS:
Behavioral: Ca CBT — Clients in intervention group will receive a CBT intervention using a manual. Intervention was developed for use in primary and secondary care using a series of qualitative studies (Naeem et al a, 2010, Naeem et al c, 2009, Naeem et al, 2009, Naeem et al, in press) during the last 5 years in Pakistan and has proven to be effective in a pilot study (Naeem et al, 2011). Intervention will consist of 6 sessions and will focus on psycho-education, symptoms management, changing negative thinking, problem solving, improving relationships and communication skills. One person from the family will be involved as a facilitator.
  Other Names: Culturally adapted Brief Cognitive Behaviour Therapy
  Arms: Ca CBT

SUMMARY:
Cognitive behaviour therapy (CBT) has an effective evidence base in the west and is recommended by the national bodies in many countries in the West. Our group has adapted CBT for depression and psychosis in Pakistan for use with local clients. Initial evaluations have found that these therapies are effective. However, due to the financial restraints it would be useful if the investigators find that brief version of the CBT might be applicable and effective in non western cultures. Therefore in this study, the investigators will be testing effectiveness of brief version of culturally adapted CBT for depression in a randomized controlled trial (RCT) in Pakistan.

DETAILED DESCRIPTION:
BACKGROUND There is a strong evidence base in favour of the CBT on its role in treating Depression and Anxiety (Embling et. al., 2002; Thase et. al., 2000; Rief. et .al, 2000)). CBT has been shown to be effective for prophylaxis (Shaw, 1989) and for the prevention of depressive relapse (Paykel et al, 1999, Fava et al; 1999). The current evidence suggests that Cognitive Behaviour Therapy (CBT) is as effective as antidepressants for treating depression (DeRubeis, Hollon et al. 1982; Murphy, Simons et al. 1984; Simons, Murphy et al. 1986), and is more effective than antidepressants in preventing relapse (Evans, Hollon et al. 1992; Hollon, DeRubeis et al. 1992). CBT is now included in national treatment guidelines in the USA and the UK (e.g. APA, 2004; NICE, 2004). However, in spite of the large body of the evidence suggesting effectiveness of the CBT for depression in the West, little progress has been made in its delivery in developing countries.

Cognitive behavioral therapy for depression was developed by Beck (Beck et al, 1979). CBT focuses on "how depressed people think and perceive themselves, others and their future". The key aspects of therapy include, taking an educative approach, working in collaboration with the client and develop insights through a Socratic dialogue. The therapist helps the depressed person to learn to recognize his "negative thinking patterns" and to re-evaluate his thinking. Clients are asked to carry out exercises at home to learn new ways of dealing with their problems (called homework). Modern psychotherapies were developed in the west and hence are likely to be underpinned by western values. It is therefore believed that CBT might need modification before it can be used in the non-western cultures because it involves exploration and attempts to modify automatic thoughts and core beliefs (Padesky et al, 1995). A systematic literature search found few studies of cognitive therapy from the non western world. However, the research so far indicates towards effectiveness of this therapy (Sumathipala, 2008, Araya et al, 2003, Wong et al, 2008 & Rahman et al, 2009). We have adapted CBT for depression in Pakistan (Naeem et al, 2009) and a pilot study to evaluate the effectiveness of CBT has shown it to be effective (Naeem et al, 2011).

The focus of the mental health services in Pakistan seem to be in the secondary care. Psychiatric services are available in major cities and patients come to see professionals from around the country. As such it seems only logical that we try to assess the effectiveness of CBT in secondary care. However, given the deficits in resources both human and financial, as well as based on the experience of our team, it will make more sense if we evaluate brief interventions. In this trial we would like to test the applicability of a brief culturally adapted CBT for patients with depression who attend secondary care in Pakistan.

Methodology Objective To assess effectiveness of brief Culturally Sensitive CBT (CS-CBT) for depression against care as usual.

Study design and duration This study is a Randomized Control Trial (RCT) which aims to assess effectiveness of brief Culturally Sensitive CBT (CS-CBT) against care as usual for depression. Study participants will be randomly assigned to two groups the intervention group will receive brief CBT developed and adapted for use in Pakistan using a series of qualitative studies (Naeem et.al 2009).

Intervention focuses on psycho-education, symptoms management, changing negative thinking, behavioral activation, problem solving, improving relationships and communication skills. One person from the family will be involved in order to improve compliance with therapy and follow up. The intervention consists of 6 sessions, plus one additional session for family.

The assessments will be carried out at the base line and then at the end of therapy (8 weeks). Control group will receive care as usual. In Pakistan this usually means, contact with a medical professional and being on antidepressants. A number equal to intervention group will be employed in this group. Bind raters will be used to assess the change in depression.

Inclusion and exclusion criteria All those who fulfill the diagnostic criteria of Depressive episode (F32) or Recurrent depressive disorder (F33 except 33.4 ) using ICD10 RDC (based on interviews using SCAN Urdu version), are between the ages of 18-60, score 8 or more on HADS, Depression Subscale, and who live within traveling distance of the psychiatry department will be approached. Those patients, who have agreed to enter the study, will be assessed 2 weeks later, to fill in the baseline measures when they attend their first appointment. Patients will be asked to attend a further appointment at the end of study period and will be assessed again.

The exclusion criteria include; excessive use of alcohol or drugs (using ICD 10 RDC for alcohol or drug abuse or dependence) significant cognitive impairment (for example learning disability or dementia) and active psychosis.

Procedure Patients who have been referred for the study will be provided brief information about the study. Those who meet the criteria and consent will be then asked to join the study and will be allocated to one arm of the trial after randomization.

Sample size Based on our pilot study, we calculated sample size for larger trial based on comparison between groups in terms of the change in the HADS Depression scores. A difference of 2 units between groups would be of clinical importance. Pilot data suggests that the within group standard deviation of the change in values over time is 3 units. With a 5% significance level and 90% power it is calculated that 48 subjects per group are required, 96 in total. It is expected that up to 30% of patients will drop out of the study. To allow for this it is planned to recruit 140 subjects into the study.

Randomization Randomization will be performed distantly by a statistician, from the list of all the patients who have been accepted for each group. After randomization patients will be allocated to either treatment or the control arm. Randomization will be performed for each group separately.

INSTRUMENTS The Bradford Somatic Inventory (BSI) (Mumford et al, 1991) is used to measure somatic symptoms. An Urdu version is available. It was developed in South Asia. It has been widely used. It has 45 items. Scores above 21 indicate depression. It was developed from symptom reports by psychiatric patients in Pakistan and Britain with clinical diagnoses of anxiety or depression. The BSI inquires about a wide range of somatic symptoms during the previous month, and if the subject has experienced a particular symptom, whether the symptom has occurred on more or less than 15 days during the month (scoring 2 or 1, respectively).

The Hospital Anxiety and Depression Scale (HAD) (Zigmond and Snaith, 1983) is a 14 item, self assessment scale designed to measure anxiety and depression. It has a high internal consistency, face validity and concurrent validity. Even-numbered questions relate to depression and odd-numbered questions relate to anxiety. Each question has 4 possible responses. Responses are scored on a scale from 3 to 0. The maximum score is therefore 21 for depression and 21 for anxiety. A score of 11 or higher indicates the probable presence of the mood disorder with a score of 8 to 10 being just suggestive of the presence of the respective state. The two subscales, anxiety and depression, have been found to be independent measures. In its current form the HADS is now divided into four ranges: normal (0-7), mild (8-10), moderate (11-15) and severe (16-21).

Brief Disability Questionnaire (BDQ) was developed by the WHO to measure disability due to physical and psychological problems and has been used extensively in research (Von Korff et al., 1996).

A data form will be used to collect information from the client.

Study sites Trial will be carried out in psychiatry departments in Lahore/Karachi, Pakistan Acknowledgements We will acknowledge the psychology graduates, R&D, LIRD and PACT for their support in publications.

INTERVENTION Clients in intervention group will receive a CBT intervention using a manual. Intervention was developed for use in primary and secondary care using a series of qualitative studies (Naeem et al a, 2010, Naeem et al c, 2009, Naeem et al, 2009, Naeem et al, in press) during the last 5 years in Pakistan and has proven to be effective in a pilot study (Naeem et al, 2011). Intervention will consist of 6 sessions and will focus on psycho-education, symptoms management, changing negative thinking, problem solving, improving relationships and communication skills. One person from the family will be involved as a facilitator.

Withdrawals and dropouts During our work in Pakistan to modify CBT for use in Pakistan, we have noticed that patients frequently drop out of therapy. We have incorporated techniques to address this issue in therapy manual, which improved drop out rates. These include giving the patients a direct number (can be a mobile phone or a wireless phone), contacting them once or twice a week to remind them of their homework and to attend the follow up sessions, speaking in client's language with minimum number of English terms and establishing a good rapport and a trusting relationship during the session. However, the risk of dropout remains high. Therefore, we will employ a higher number of clients in our study, with a probable dropout rate of 30%.

Data entry and analysis Statistical analyses would be carried out using an intention to treat. Analyses will be carried out using SPSS v16 . Both parametric and non parametric tests will be carried out as appropriate to compare groups. An analysis of covariance will be used to measure the differences between the two groups at three time points, where the data is normally distributed. A t test will be used to compare groups, both paired and unpaired. SPSS frequency and descriptive commands will be used to measure descriptive statistics. SPSS explore command will be used to measure normality of the data, using histograms and Kolmorogov Smirnov test. If the therapy is proved to be more effective than the control, we will also use a binary logistic regression analysis to explore factors which predict good outcome. An intention to treat analysis will be performed. Number Needed to Treat (NNT) will be calculated to assist clinicians with clinical decision making.

Research in clinically naturalistic settings It is recognized that such research is most likely to provide results that are relevant to routine clinical practice; the current study provides a more rigorous evaluation for an intervention that can be provided in current service in Pakistan and at no extra costs.

ELIGIBILITY:
Inclusion Criteria:

* All those who fulfil the diagnostic criteria of Depressive episode (F32) or Recurrent depressive disorder (F33 except 33.4 ) using ICD10 RDC (based on interviews using SCAN Urdu version),
* Are between the ages of 19-60,
* Score 8 or more on HADS, Depression Subscale, and
* Who live within traveling distance of the psychiatry department will be approached

Exclusion Criteria:

* Excessive use of alcohol or drugs (using ICD 10 RDC for alcohol or drug abuse or dependence)
* Significant cognitive impairment (for example learning disability or dementia) and
* Active psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and depression Rating Scale- Depression subscale | Participants will be assessed at baseline and then end of therapy at 12 weeks
  Measurement of depression

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale, Anxiety subscale | Participants will be assessed at baseline and then end of therapy at 12 weeks
  Measurement of anxiety
Bradford Somatic Inventory | Participants will be assessed at baseline and then end of therapy at 12 weeks
  Measurement of somatic symptoms
Brief disability questionnaire | Participants will be assessed at baseline and then end of therapy at 12 weeks
  To measure disability associated with depression

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, MRCPsych,PhD, Principal Investigator — Pakistan Association of Cognitive Therapists
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Pakistan